CLINICAL TRIAL: NCT03370575
Title: A Randomized, the Second-generation Non-ionic Monomer Contrast Parallel Control, Multicenter Clinical Study to Evaluate the Imaging Diagnostic Quality and Fertility Promoting Effect of Ethiodized Poppyseed Oil in Hysterosalpingography of Infertile Patients.
Brief Title: RCT of Ethiodized Poppyseed Oil VS the Second-generation Non-ionic Monomer Contrast in Hysterosalpingography of Infertile Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jing zhang, Director of medical imaging, Guangzhou Women and Children's Medical Center, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017102708
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ethiodized poppyseed oil (Experimental)
  Interventions: Drug: ethiodized poppyseed oil
- the second-generation non-ionic monomer contrast (Active Comparator)
  Interventions: Drug: the second-generation non-ionic monomer contrast

INTERVENTIONS:
Drug: ethiodized poppyseed oil — Hysterosalpingography using ethiodized poppyseed oil
  Arms: ethiodized poppyseed oil
Drug: the second-generation non-ionic monomer contrast — Hysterosalpingography using the second-generation non-ionic monomer contrast
  Arms: the second-generation non-ionic monomer contrast

SUMMARY:
This study evaluates the difference of imaging diagnostic quality and fertility promoting effect in the diagnosis and treatment of infertility by hysterosalpingography between using ethiodized poppyseed oil and the second-generation non-ionic monomer contrast. Half of participants will receive ethiodized poppyseed oil for hysterosalpingography, while the other half will receive the second-generation non-ionic monomer contrast for hysterosalpingography.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 to 39 years, Female;
* Had spontaneous menstrual cycle;
* Had been trying to conceive for at least 1 year;
* There was an indication for evaluation of tubal patency by means of hysterosalpingography.
* Understand and sign informed consent.

Exclusion Criteria:

* Known endocrine disorders(e.g., the polycystic ovary syndrome, diabetes, hyperthyroidism, and hyperprolactinemia);
* Less than eight menstrual cycles per year;
* A high risk of tubal disease (as indicated by a history of pelvic inflammatory disease, previous chlamydia infection, or known endometriosis);
* Hyperthyroidism;
* Vaginitis, acute or subacute pelvic inflammatory active phase, uterus or fallopian tube tuberculosis;
* Uterine or cervical bleeding;
* Menelipsis without excluding pregnancy;
* Severe heart disease and lung disease;
* Body temperature beyond 37.5 ℃ within 3 days before hysterosalpingography;
* A total motile sperm count of <1 million sperm per milliliter;
* Complications or social environment that can cause patients to fail to follow the study plan and even endanger the patient's safety.

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Imaging diagnostic quality of hysterosalpingography | procedure (during hysterosalpingography)
  defined as mean scores of 3 pictures shot at certain points
Ongoing pregnancy | 15 months （6 months for recruitment, 9 months for ongoing pregnancy）
  defined as the first day of the last menstrual cycle for the pregnancy is within 6 months after randomization, and after 12 weeks of gestation a positive fetal heartbeat is on ultrasonographic examination

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (13):
- China (13):
  - Beijing Haidian District Maternal and Child Care Service Centre, Beijing, Beijing Municipality
  - The second affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangzhou women and children's medical center, Guangzhou, Guangdong
  - Liuzhou Maternal and Child Care Service Centre, Liuchow, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Maternal and Child Care Service Centre, Wuhan, Hubei
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Lianyungang Maternal and Child Care Service Centre, Lianyungang, Jiangsu
  - Nanjing Maternal and Child Care Service Centre, Nanjing, Jiangsu
  - Dalian Women and Children Medical Center, Dalian, Liaoning
  - Fudan University affiliated Maternity Hospital, Shanghai, Shanghai Municipality
  - Jinjiang Maternal and Child Care Service Centre, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Zhang J, Lan W, Wang Y, Chen K, Zhang G, Yang W, Chen H, Xu W, Ma J, Qin W, Zhang Y, Wang W, Wang H, Dong Z, Wang Y, Chen Y, Gang N, Tang Y. Ethiodized poppyseed oil-based contrast medium is superior to water-based contrast medium during hysterosalpingography regarding image quality improvement and fertility enhancement: A multicentric, randomized and controlled trial. EClinicalMedicine. 2022 Apr 5;46:101363. doi: 10.1016/j.eclinm.2022.101363. eCollection 2022 Apr. PMID 35399811